CLINICAL TRIAL: NCT00076804
Title: DOT-HAART for HIV-Infected South African Adults
Brief Title: Helping HIV Infected Patients in South Africa Adhere to Drug Regimens
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB stopped trial for futility
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Dr. Richard Chaisson, Director, Center for TB Research, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI055359-01A1 (NIH); 1R01AI055359-01A1 (NIH)
Record Dates: First submitted 2004-02-03; First posted 2004-02-06 (Estimated); Results first posted 2010-07-02 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: Directly Observed Therapy; DOT
MeSH Terms: conditions — HIV Infections; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Use of a patient nominated peer supporter who will observe the morning dose of ARVs
  Interventions: Behavioral: Directly Observed Therapy
- 2 (No Intervention): Self administration of ARVs

INTERVENTIONS:
Behavioral: Directly Observed Therapy — Use of a patient nominated peer supporter who will observe the morning dose of ARVs
  Arms: 1

SUMMARY:
Three or more anti-HIV drugs are taken in combination as part of a treatment regimen. These drug regimens must be closely followed in order to be successful. Having a support person watch a patient take his or her anti-HIV drugs each day may help a patient follow his or her regimen. This study will see if patient-chosen treatment supporters help patients take HIV medicines correctly and improve their health.

Study hypothesis: The mean change in CD4 count at 12 and 24 months will be significantly higher in the directly observed therapy-highly active antiretroviral therapy (DOT-HAART) arm as compared to the self-administered arm.

DETAILED DESCRIPTION:
South Africa has one of the worst and fastest growing HIV epidemics in the world. Highly active antiretroviral therapy (HAART) has been shown both at the individual and public health levels to reduce morbidity, mortality, and vertical and possibly horizontal HIV transmission. However, expenses, feasibility, long-term adherence, and effective delivery of HAART remain formidable barriers, particularly in developing nations. Recently, international initiatives have provided hope for widespread use of HAART at affordable cost in sub-Saharan Africa. Simplified, once-daily HAART regimens with directly observed therapy (DOT) may help to achieve high levels of treatment adherence, a key component for long-term viral suppression and treatment success. Peer advocates have been used to improve adherence with medical therapies in a variety of settings. This study will evaluate the effectiveness and feasibility of DOT using patient-nominated peer supervisors to improve adherence to HAART in HIV infected adults in South Africa.

Participants will be randomly assigned to either Peer-DOT-HAART or self-administration of a once-daily combination of the Western Cape Province ART program medications for 24 months. Study measures will include CD4 cell count and HIV viral load, adherence questionnaires, genotypic HAART resistance testing, and incidence of new or recurrent opportunistic infections.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Viral load greater than 1000 copies/ml
* CD4 count of 200 cells/mm3 or less, or World Health Organization Stage 4 disease
* Living in the area of the study site
* Had a known address for more than 3 months
* Willing to nominate a treatment supervisor (a close family member, sexual partner, friend, or community volunteer) to observe daily ingestion of tablets
* Willing to disclose HIV status to a treatment supervisor and ready to commit to long-term antiretroviral therapy
* Acceptable methods of contraception

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Chaisson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- University of Cape Town, Cape Town, South Africa

REFERENCES:
- [Result] Nachega JB, Chaisson RE, Goliath R, Efron A, Chaudhary MA, Ram M, Morroni C, Schoeman H, Knowlton AR, Maartens G. Randomized controlled trial of trained patient-nominated treatment supporters providing partial directly observed antiretroviral therapy. AIDS. 2010 Jun 1;24(9):1273-80. doi: 10.1097/QAD.0b013e328339e20e. PMID 20453627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study site was a public sector ART clinic at the GF Jooste Hospital, a secondary level facility in Cape Town, Western Cape province of South Africa, serving several peri-urban townships. Enrollment began February 13, 2005, and ended on July 7, 2007, with the last follow-up occurring on July 25, 2008.
Groups:
- Peer Supporter: Use of a patient nominated peer supporter who sill observe the morning dose of ARVs
- Self Administration: Self administration of ARVs
Period: Overall Study
Arm/Group | Peer Supporter | Self Administration
Started | 137 | 137
Completed | 77 (111 completed week 48, 77 completed week 96.) | 68 (102 completed week 48, 68 completed week 96)
Not Completed | 60 | 69
Not completed — Death | 9 | 20
Not completed — Lost to Follow-up | 9 | 9
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Early study Closure | 32 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Supporter | Self Administration | Total
Number analyzed (Participants) | 137 | 137 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 136 | 270
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (9.7) | 36.7 (9.2) | 36.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 58 | 58 | 116
Region of Enrollment [Number; unit: participants]
  South Africa | 137 | 137 | 274

OUTCOME MEASURES:

1. Primary Outcome: Impact of DOT Compared to Self-administered Treatment as Measured by HIV Viral Load at 12 Months of Treatment
Description: Proportion of Patients with HIV RNA Levels of <400 at 12 Months - Intention-to-treat
Time Frame: at 12 and 24 months of treatment
Measure: Number; unit: participants
Arm/Group | Peer Supporter | Self Administration
Number analyzed (Participants) | 136 | 136
participants | 99 | 93
Statistical Analysis 1: Comparison: Peer Supporter vs Self Administration; Unadjusted endpoint analyses were conducted on an intention-to-treat basis using all patients enrolled to compare outcomes in the DOT vs. Self-ART arm. For viral load analyses, missing values were considered detectable (missing¼failure analysis). As-treated analyses were also conducted using patients remaining in the study with available data.Crosssectional comparisons between study groups were conducted using two sample t-test,Wilcoxon rank-sum test,chi-squared orFisher's exact and Kaplan-Meier; Test type: Superiority or Other; p = 0.42, Chi-squared — Logistic regression analysis & Cox proportional hazards regression analyses were performed to compare outcomes after adjusting for the relevant covariates,including study arm, age, sex, baseline CD4 cell counts and viral load and pill count adherence; one degree of freedom

2. Primary Outcome: Impact of DOT Compared to Self-administered Treatment as Measured by HIV Viral Load at 24 Months of Treatment
Description: Proportion of Patients with HIV RNA Levels of <400 Copies/mL at 24 Months [Intention-to-treat (ITT)
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Peer Supporter | Self Administration
Number analyzed (Participants) | 104 | 104
participants | 63 | 62
Statistical Analysis 1: Comparison: Peer Supporter vs Self Administration; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.89, Chi-squared — [p-value comment as in outcome 1, analysis 1]; one degree of freedom

3. Primary Outcome: Immunological Response: Median CD4 (IQR) Cell Count Increase From Baseline at 12 Months by Study Arm
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | Peer Supporter | Self Administration
Number analyzed (Participants) | 105 | 100
cells/uL | 185 [108 to 276] | 160 [78 to 236]
Statistical Analysis 1: Comparison: Peer Supporter vs Self Administration; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Immunological Response: Median CD4 (IQR) Cell Count Increase From Baseline at 24 Months by Study Arm
Time Frame: 24 months
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | Peer Supporter | Self Administration
Number analyzed (Participants) | 84 | 77
cells/uL | 281 [144 to 403] | 262 [149 to 363]
Statistical Analysis 1: Comparison: Peer Supporter vs Self Administration; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected throughout the duration of the study. It was assessed at each clinic visit and if the subject presented between visits.
Arm/Group | Peer Supporter | Self Administration
Serious Adverse Events (participants affected / at risk) | 19/137 | 29/137
Other Adverse Events (participants affected / at risk) | 71/137 | 89/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Supporter (N=137) | Self Administration (N=137)
Death (General disorders) | 9 (9) | 20 (20)
DAIDS Grade IV AE (General disorders) | 5 (5) | 2 (2)
Hospitalization (General disorders) | 5 (5) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Supporter (N=137) | Self Administration (N=137)
AIDS-Defining Illness (General disorders) | 22 (28) | 31 (35)
DAIDS Grade III Event (General disorders) | 17 (22) | 21 (25)
New Diagnosis/Worsening Medical Condition (General disorders) | 32 (39) | 37 (52)

LIMITATIONS AND CAVEATS:
Intervention was stopped at 12 months, transition phase did not ensure that participants developed a set of adherence strategies to replace DOT-ART. Low incidence of AIDS-defining illness and death limit our ability to make final conclusions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No